CLINICAL TRIAL: NCT03646669
Title: Symptom Perception, Behavior, and Outcomes in Older Asthmatics
Brief Title: Symptom Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Albert Einstein College of Medicine (Other); Jacobi Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan P Wisnivesky, Professor of Medicine and Chief, Division of General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 15-0667; R01HL131418 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Older adults; Asthma; Symptom perception; Self-management behaviors; Medication adherence
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma education and PEF feedback (Experimental): Patients receive asthma education and personal Peak expiratory flow (PEF) feedback
  Interventions: Behavioral: PEF Feedback
- Asthma education (Placebo Comparator): No PEF feedback arm
  Interventions: Behavioral: Asthma education

INTERVENTIONS:
Behavioral: PEF Feedback — Patients in the PEF feedback arm will receive a one-time session including asthma management education, discussion of their asthma symptoms, review of individual PEF results and perception of symptoms, and problem-solving techniques to improve asthma self-management. After the session, the participants in this arm will be able to view in the display of the AM2 device their PEF values and will be instructed to mentally note their actual results with their pre-effort estimated BPF. They will also set a motivational message for themselves that will appear on the device.
  Other Names: Intervention Arm
  Arms: Asthma education and PEF feedback
Behavioral: Asthma education — General asthma education, AM2 training, and positive counseling, but no discussion linking asthma symptom perception to SMB. Following the session, these participants will use the AM2 to track PEF actual and perceived values twice per day, but they will be blinded to the actual PEF values. Control arm patients will see a standard motivational message appear on the screen of the AM2 device.
  Arms: Asthma education

SUMMARY:
Older asthmatics have considerably worse outcomes than younger patients with asthma. In this study, the investigators will evaluate the role of symptom perception as a key determinant of poorer outcomes and lower adherence to asthma self-management behaviors among older asthmatics. The proposed study is significant for its potential to greatly advance understanding of the mechanisms related to worse outcomes in older adults, and it will provide actionable data for new interventions to improve self-management.

DETAILED DESCRIPTION:
Asthma is a common condition in the older population and associated with worse morbidity and mortality compared to younger individuals. Various self-management behaviors (SMB), medication adherence in particular, are key for achieving good asthma control. Unfortunately, less than half of older asthmatics regularly adhere to their controller medications and to other SMB. Several observations suggest that symptom perception may be a major determinant of asthma SMB and outcomes in older adults. First, experimental studies consistently demonstrate that many older adults are substantially less aware of their level of airway obstruction. Second, under-perception of asthma symptoms is linked to elevated risk of near-fatal and fatal asthma attacks and increased morbidity among younger adults. Third, cognitive impairment, commonly associated with aging, has been identified as a key determinant of under-perception of symptoms in younger asthmatics. Fourth, interventions to correct symptom under-perception in children have been shown to improve asthma medication adherence. Despite the greater vulnerability of older asthmatics to poor asthma outcomes and their diminished ability to perceive the severity of their airway obstruction, the association of symptom perception with asthma SMB and outcomes has not been studied in this population. The goal of this project is to determine how symptom perception influences the management and outcomes of older asthmatics and to pilot test an intervention to correct under-perception. The Specific Aims are: 1) Prospectively assess the association between symptom perception and asthma morbidity among older adults; 2) Examine the association between symptom perception and asthma SMB among older adults and identify the pathways (via illness and medication beliefs) linking them; 3) Determine the influence of cognition on symptom perception among older adults with asthma; 4) Pilot test an intervention to correct under-perceptions of asthma symptoms in older adults. The investigators will conduct a prospective cohort study of 400 asthmatics ≥60 years of age recruited from East Harlem and the Bronx in New York City. The investigators will measure symptom perception in naturalistic settings using an innovative and validated methodology and repeatedly collect data on illness and medication beliefs, cognitive functioning, SMB (including objective measures of medication adherence), and asthma morbidity over 12 months. At the end of the observation period, the investigators will pilot test an intervention to improve symptom perception on a random sample of 80 participants. The proposed study is significant for its potential to greatly advance understanding of the mechanisms related to low adherence to SMB and worse outcomes in older asthmatics, a vulnerable and understudied population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* English or Spanish speaking
* Asthma diagnosis made by a health care provider

Exclusion Criteria:

* Diagnosis of dementia
* Diagnosis of chronic obstructive pulmonary disease (COPD) or other chronic respiratory illness
* Smoking history of ≥15 pack-years owing to possible undiagnosed COPD
* Moderate or severe cardiac disease (including New York Heart Association stages 4 or 5 congestive heart failure, because dyspnea among patients with severe heart failure is more likely to be attributable to their heart condition than their asthma)
* Dependence on assistance for medication administration
* Uncorrectable visual impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wisnivesky, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Albert Einstein College of Medicine/Yeshiva University, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Started | 33 | 25
Completed | 28 | 25
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma Education and PEF Feedback | Asthma Education | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (4.9) | 65.7 (5.6) | 66.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 9 | 6 | 15
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 1 | 2 | 3
Education [Count of Participants; unit: Participants]
  Less than high school | 5 | 3 | 8
  High school graduate | 5 | 2 | 7
  Some college | 8 | 9 | 17
  College graduate or higher degree | 9 | 11 | 20
  Unknown or Not reported | 1 | 0 | 1
Monthly Income [Count of Participants; unit: Participants]
  ≤$1500 | 13 | 12 | 25
  >$1500 | 12 | 10 | 22
  Unknown or Not reported | 3 | 3 | 6
Marital Status [Count of Participants; unit: Participants]
  Married | 13 | 4 | 17
  Single/Divorced/Widowed | 14 | 21 | 35
  Unknown or Not reported | 1 | 0 | 1
Health Insurance [Count of Participants; unit: Participants]
  Medicaid or Medicare | 20 | 16 | 36
  Private or Other | 6 | 6 | 12
  No insurance | 1 | 0 | 1
  Unknown or Not reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ)
Description: Change in self-reported asthma control validated survey, with a total score range from 0-6, with a higher score indicating severely uncontrolled asthma , used to assess current asthma control at pre-intervention, 1week post-pilot follow up visit and 4 weeks post-pilot follow-up visit
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 1.2 (1.1) | 1.4 (1.0)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 0.8 (0.8) | 1.4 (0.8)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 0.6 (0.5) | 1.6 (0.9)

2. Primary Outcome: Change in Asthma Quality of Life Questionnaire (AQLQ)
Description: Change in self-reported asthma-related quality of life validated survey used to assess asthma-related quality of life at at pre-intervention, 1week post-pilot follow up visit and 4 weeks post-pilot follow-up visit. Total Score from 1-7, with higher score indicating better quality of life.
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 5.2 (1.2) | 5.0 (1.0)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 5.6 (1.4) | 4.9 (1.1)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 5.7 (1.1) | 5.0 (1.1)

3. Secondary Outcome: Change in Medication Adherence Rating Scale (MARS)
Description: MARS is a self-reported questionnaire with the total score range from 0-10 with a higher score indicating better adherence.
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 4.0 (1.0) | 4.2 (0.8)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 4.4 (0.7) | 4.3 (0.8)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 4.2 (0.6) | 4.4 (0.6)

4. Secondary Outcome: Change in Beliefs About Medicines Questionnaire (BMQ) - Necessity Score and Concerns Score
Description: 10-item scale that measures beliefs about asthma controller medication in 2 subdomains: necessity and concerns. All items have a ﬁve-point Likert answer option, ranging from 1 = strongly disagree to 5 = strongly agree, with total range from 10 to 50, with higher scores indicate stronger beliefs about the corresponding concepts.
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Necessity Baseline | 17.4 (4.9) | 18.2 (4.4)
  Necessity 1 week follow up: number analyzed (Participants) | 28 | 22
  Necessity 1 week follow up | 18.9 (4.3) | 17.2 (4.5)
  Necessity 1 month follow up: number analyzed (Participants) | 28 | 22
  Necessity 1 month follow up | 18.4 (4.5) | 18.1 (5.2)
  Concerns Baseline | 14.2 (4.2) | 14.5 (4.0)
  Concerns 1 week follow up: number analyzed (Participants) | 28 | 22
  Concerns 1 week follow up | 13.0 (4.4) | 12.9 (4.5)
  Concerns 1 month follow up: number analyzed (Participants) | 28 | 22
  Concerns 1 month follow up | 13.6 (4.2) | 12.8 (4.0)

5. Secondary Outcome: Change in Beliefs About Illness Perception Questionnaire (BIPQ)
Description: The BIPQ includes 9 items designed to rapidly assess the cognitive and emotional representations of illness- consequences, timeline, personal control, treatment control, experience symptoms, concerns, emotions and comprehensibility. For analyses, the first 8 items are summed and item 9 which is part of the causal scale is excluded. Items for personal control, treatment control and comprehensibility were reverse coded. All of the 8 items, are rated using a 0 (none) to 10 (extreme) response scale giving a sum total score of 0-80. Higher total scores indicate worse asthma perception.
Time Frame: Baseline, 1 week follow up
Population: data not available for participants with missing questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 33.3 (13.9) | 34.0 (0.7)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 30.7 (13.9) | 34.7 (11.8)

6. Secondary Outcome: Symptom Perception Measures Adjusted
Description: Assessed based on alignment of patient guesses and actual PEF values recorded by the AM2 device and then categorizing into accurate, under or over-perception, adjusted for age, sex, race, monthly income Assesses if training and feedback can improve under perception of airflow obstruction and lead to better control in older adults with asthma
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
percent
  Symptom Accurate Perception Baseline | 55.3 (6.5) | 51.1 (6.9)
  Symptom Accurate Perception 1 week follow up: number analyzed (Participants) | 28 | 22
  Symptom Accurate Perception 1 week follow up | 71.5 (6.3) | 52.7 (6.4)
  Symptom Accurate Perception 1 month follow up: number analyzed (Participants) | 28 | 22
  Symptom Accurate Perception 1 month follow up | 72.2 (7.6) | 42.9 (8.3)
  Symptom Under-Perception Baseline | 39.7 (7) | 44.9 (7.5)
  Symptom Under-Perception 1 week follow up: number analyzed (Participants) | 28 | 22
  Symptom Under-Perception 1 week follow up | 11.9 (6.4) | 33.8 (6.4)
  Symptom Under-Perception 1 month follow up: number analyzed (Participants) | 28 | 22
  Symptom Under-Perception 1 month follow up | 11.8 (7.4) | 45.1 (8.0)
  Symptom Over-Perception Baseline | 5.0 (2.1) | 3.9 (2.3)
  Symptom Over-Perception 1 week follow up: number analyzed (Participants) | 28 | 22
  Symptom Over-Perception 1 week follow up | 16.6 (4.9) | 13.6 (5)
  Symptom Over-Perception 1 month follow up: number analyzed (Participants) | 28 | 22
  Symptom Over-Perception 1 month follow up | 16 (5.9) | 12 (6.4)
  Actual Best, personal best baseline | 67 (0.4) | 68.2 (0.6)
  Actual Best, personal best 1 week follow up | 80.8 (0.6) | 71.9 (0.7)
  Actual Best, personal best 1 month follow up | 78.6 (0.5) | 67.7 (0.7)

7. Secondary Outcome: Asthma Control Questionnaire (ACQ) Score - Adjusted
Description: Change in self-reported asthma control validated survey, with a total score range from 0-6, with a higher score indicating severely uncontrolled asthma, used to assess current asthma control at pre-intervention, 1week post-pilot follow up visit and 4 weeks post-pilot follow-up visit adjusted for age, sex, race, monthly income
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 1.4 (0.2) | 1.5 (0.2)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 0.9 (0.4) | 1.1 (0.4)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 0.7 (0.3) | 1.3 (0.3)

8. Secondary Outcome: Treatment Credibility
Description: Treatment Credibility adjusted for age, sex, race, monthly income
  The credibility of a treatment rationale consists of "how believable, convincing, and logical the treatment is". The CEQ credibility factor, reflecting a cognitively-based process, is based on patients' summed responses to three items measuring how logical the therapy seems, how successful one thinks it will be in reducing symptoms, and how confident one would be in recommending it to a friend with similar symptoms. The modified version used in this study included items rated on 7 point scales ranging from 1 (Not at all logical/successful /confident) to 7 (Very logical/successful /confident), with a total score possible range of 3 to 21. Higher scores indicate higher treatment credibility.
Time Frame: 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 19.3 (1.7) | 19.2 (1.5)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 19.2 (1.4) | 18.9 (3.7)

9. Secondary Outcome: Treatment Expectancy
Description: Treatment Expectancy adjusted for age, sex, race, monthly income.
  Outcome expectancy consists of patients' beliefs about how likely they are to benefit from a treatment.
  The CEQ expectancy factor, reflecting an affectively-based process, is based on patients' responses to three items reflecting how much they think they will improve by the end of treatment, how much they feel therapy will help reduce their symptoms, and how much they feel they will improve by the end of treatment. Because one item is on the same 7-point scale as the credibility items and two are assessed on an 11-point scale (from 0% to 100% in 10-point increments), responses are first standardized before summing to render the expectancy total score. The total score possible range is 3 to 33. Higher scores indicate higher treatment expectancy.
Time Frame: 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  1 week follow up | 25.3 (4.6) | 25.2 (2.7)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 25.3 (4.8) | 21.9 (8.9)

10. Secondary Outcome: Change in Medication Adherence Rating Scale (MARS) Adjusted
Description: MARS is a self-reported questionnaire with the total score range from 0-10 with a higher score indicating better adherence. MARS, adjusted for age, sex, race, monthly income
Time Frame: Baseline, 1 week follow up, 1 month follow up
Population: data not available for participants with missing questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
Number analyzed (Participants) | 28 | 25
score on a scale
  Baseline | 4.0 (0.2) | 4.3 (0.2)
  1 week follow up: number analyzed (Participants) | 28 | 22
  1 week follow up | 4.4 (0.2) | 4.2 (0.2)
  1 month follow up: number analyzed (Participants) | 28 | 22
  1 month follow up | 4.1 (0.1) | 4.4 (0.2)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Asthma Education and PEF Feedback | Asthma Education
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03646669/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03646669/SAP_001.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03646669/ICF_002.pdf